CLINICAL TRIAL: NCT04223440
Title: Ultrasonographic and MRI Explorations of Infraspinatus Muscle in Postero-superior Rotator Cuff Tear
Acronym: VISUMIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DR190044
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Tears; MRI; Ultrasonographic explorations
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postero-superior Rotator Cuff Tear (Experimental): MRI, ultrasonographic explorations
  Interventions: Other: MRI; Other: ultrasonographic explorations
- Healthy Postero-superior Rotator Cuff (Other): MRI, ultrasonographic explorations
  Interventions: Other: MRI; Other: ultrasonographic explorations

INTERVENTIONS:
Other: MRI — MRI on both shoulder
Other: ultrasonographic explorations — ultrasound and elastography explorations on both shoulder

SUMMARY:
The project aims to evaluate the contribution of texture analysis on MRI sections, and the technical feasibility, reproducibility, and clinical relevance of quantitative ultrasound and elastography to characterize the composition and volume of infraspinatus muscle in postero-superior rotator cuff tears. The perspectives are to optimize the imaging to allow a quantitative, objective and reproducible analysis of the muscle tissue and its characteristics.

DETAILED DESCRIPTION:
The rotator cuff of the shoulder consists of 4 tendinomuscular units including the infraspinatus. This complex system fulfils a double role: stabilization/coaptation (raising the arm) and arm mobility (especially external rotation). Rupture of rotator cuff tendons is frequent (> 80% among chronic shoulder pain). They go with a decrease in muscle volume (amyotrophy) and irreversible fat infiltration. The treatment is medical and then surgical (if necessary). The degrees of atrophy and muscle infiltration (especially infraspinatus) are the criteria of choice for surgery. Actually, they are assessed in MRI according to the classification of Fuchs; it is operator dependent, qualitative and poorly reproducible with a strong inter-observer variability. Our team highlighted (2016) the possibility of using texture analysis software to objectively measure the proportion of fatty tissue on MRI sections of the cuff rotator muscles. This work also showed the possibility of using mode B ultrasound for morphological imaging and shear wave elastography to estimate the elasticity of the infraspinatus. The project aims to evaluate the contribution of texture analysis on MRI sections, and the technical feasibility, reproducibility, and clinical relevance of quantitative ultrasound and elastography to characterize the composition and volume of infraspinatus muscle in postero-superior rotator cuff tears. The perspectives are to optimize the imaging to allow a quantitative, objective and reproducible analysis of the muscle tissue and its characteristics.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 35 years-old and ≤75 years-old
* tendonous, transfixing, postero-superior, unilateral and symptomatic rotator cuff lesions
* controlateral shoulder without symptom, without rotator cuff injuries, without medical ou surgical history
* written informed consent
* affiliation to a social security system

Exclusion Criteria:

* pregnant woman
* patient under legal protection
* contraindications to MRI
* traumatic or surgical or medical relevant history on shoulder
* general or local disease affecting the skeletal striated muscle

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
MRI Texture Index (MTI) | up to 2 months
  MRI texture index (MTI) on the healthy side and pathological side

SECONDARY OUTCOMES:
Ultrasound Texture Index (UTI) | up to 2 months
  Ultrasound Texture Index (UTI) on the healthy side and pathological side
velocity of shear wave in m.s-1 | up to 2 months
  shear wave velocity on the healthy side and pathological side

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No